CLINICAL TRIAL: NCT05458115
Title: Clinical Study of MRD Recurrence Monitoring After Surgical Resection of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: kyMRD
Record Dates: First submitted 2021-09-16; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: HCC
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver resection group
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Patient underwent hepatic R0 resection within a week

SUMMARY:
ctDNA-based liquid biopsy can better detect the presence of MRD before imaging and serological markers, and is suitable for postoperative MRD and recurrence monitoring, which has been clinically validated in several cancer types such as lung cancer and intestinal cancer. However, there is no systematic comparative study of postoperative MRD and recurrence monitoring based on ctDNA testing in hepatocellular carcinoma. A prospective multicenter observational clinical study is proposed to evaluate the use of liquid biopsy based on ctDNA NGS assay in surgical evaluation, MRD and molecular recurrence state monitoring after radical resection of hepatocellular carcinoma, and to compare with imaging and serological findings with the aim of early detection of disease recurrence or metastasis and more survival benefits for patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria.

1. understood and agreed to follow the study requirements, were willing to provide samples for testing, and signed an informed consent form.
2. age 18-75 years, regardless of gender.
3. patients with a clinical diagnosis of surgically resectable CNLC Ia-IIa hepatocellular carcinoma.
4. patients who have not received any previous treatment for their primary treatment and who agree to receive treatment
5. an ECOG physical status of 0 or 1 within 1 week prior to enrollment.
6. have at least one measurable lesion according to RECIST v1.1 or mRECIST criteria and have not received radiation therapy
7. an expected survival time of ≥ 3 months.
8. adequate organ function, with the following laboratory test values required within 7 days prior to treatment: - Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 90 g/L, and white blood cell count ≥ 3 × 109/L.

Note: Patients should not have received blood transfusion or growth factor support within 14 days prior to blood sample collection.

* International normalized ratio (INR) ≤ 1.5 times the upper limit of normal (1.5 x ULN).
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN.
* Total serum bilirubin ≤ 1.5 x ULN (patients with Gilbert syndrome may be enrolled if total bilirubin < 3 x ULN).
* Glutathione aminotransferase (AST) and glutathione alanine aminotransferase (ALT) ≤ 2.5 x ULN.
* Renal function: serum creatinine ≤ 1.5× ULN or creatinine clearance ≥ 50 mL/min according to Cockcroft-Gault formula

Exclusion Criteria:

1. patients with comorbid other active malignancies.
2. active infection or known human immunodeficiency virus infection (HIV-positive).
3. previous allogeneic stem cell transplantation.
4. the patient's compliance during the study period is, in the judgment of the investigator, inadequate
5. having received any systemic antineoplastic therapy prior to initiation of study treatment with approved
6. has received blood transfusion, radiotherapy, or drug therapy within 1 month prior to enrollment.
7. untreated active hepatitis C (patients with positive anti-HCV antibodies or positive HCV RNA cannot be enrolled); untreated active hepatitis B (HBsAg positive and HBV DNA ≥ 2000 IU/mL).
8. patients with hepatocellular carcinoma in whom distant metastases, vascular invasion and cancer emboli have been observed on imaging
9. women of childbearing age with positive blood pregnancy tests
10. subjects with a history of serious systemic disease such as diabetes, hypertension, myocardial infarction, etc., or other reasons believed to interfere with the accuracy of the test, or a combination of serious mental illness, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
clinicopathological information recording | 2 years
  Age, gender, ECOG PS, Child-pugh, tumor stage, cirrhosis, history of hepatitis
Adverse effect | 2 years
  Incidence of adverse reactions after various treatments